CLINICAL TRIAL: NCT04275011
Title: Bone Response to Resistance and Impact Exercise (BRRIE) in Women on Antiresorptive Medications: A Randomized Controlled Trial
Brief Title: Bone Response to Exercise in Women on Antiresorptive Medications
Acronym: BRRIE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been terminated
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 41153
Record Dates: First submitted 2020-02-03; First posted 2020-02-19 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Osteoporosis; Bone Loss
Keywords: Exercise; Progressive Resistance Training; Impact Exercise; Anti-resorptive medication
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a single-blinded RCT comparing moderate-high progressive resistance training and impact exercise to an attention control who will be performing static posture and balance exercises.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Using a computer-generated random selection process, participants will be randomized in a 1:1 allocation ratio in blocks which will be randomly determined. Allocation will be concealed from all but the person performing the randomization, the participants, and the exercise trainers. Although the participants cannot be blinded to the assigned exercise group, they will simply be informed that the purpose of the study is to compare two different exercise programs with no indication regarding the study hypothesis. Research staff blinded to group allocation will have access to the assessment forms. An alternate research staff member will collect or enter data that may cause unblinding (e.g., randomization, exercise adherence logs). Exercise trainers who are unblinded to group allocation will have access to the exercise training manual. Completed outcome assessments and exercise training data will be stored in separate password protected files to avoid exposing group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static Posture and Balance Exercise (Active Comparator): Participants in the control group will receive equal attention through a static posture and balance exercise class two times per week, in a small group setting.
  Interventions: Other: Static Balance and Postural Exercise
- Progressive Resistance and Impact Exercise (Experimental): The exercise program will include two progressive resistance and impact exercise training sessions per week in a small group setting. Exercises will be individually tailored to the participants' abilities and designed to achieve a maximum 80-85% 1RM.
  Interventions: Other: Progressive Resistance and Impact Exercise

INTERVENTIONS:
Other: Progressive Resistance and Impact Exercise — Full body resistance and impact exercises will be performed twice a week for 30-45 minutes over a 6 month period. There will be at least one day of rest between scheduled exercise sessions. Participants will be individually prescribed variations of push, pull, squat, lift and carry movements targeting major muscle groups that they can safely complete, and accessory exercises to help develop movement patterns. Exercises will challenge both the upper and lower body using functional movement patterns. Each muscle group will be trained twice a week. During the first month, participants will focus on completing exercises with good form at a low intensity. Once form is mastered, exercises will be progressed (by increasing load, or challenge of the movement) to a moderate to high exercise intensity (80-85% 1RM) so that the participant can complete a maximum of 8 (~80% 1RM) or 6 (~85% 1RM) repetitions with 1-2 repetitions in reserve for 3 sets at a rating of perceived exertion (RPE) of 8-9.
  Arms: Progressive Resistance and Impact Exercise
Other: Static Balance and Postural Exercise — Participants in the attention control group will perform static posture and balance exercises (e.g., low intensity yoga poses) and will be given the same attention as the participants in the intervention group. The small group exercises will be performed twice a week, 30-45 minutes per session, over 6 months, with at least one day of rest between each session. The exercise program will be supervised by a certified personal trainer and yoga instructor who is BoneFit trained.
  Arms: Static Posture and Balance Exercise

SUMMARY:
Performing resistance training and impact exercise at a moderate to high intensity may help prevent bone loss. However, medications used to treat bone diseases such as osteoporosis reduce the activity of bone cells. The investigators are unsure whether bone cells will still respond to exercise in people on osteoporosis medications. Therefore, investigators have designed a study to compare bone response to moderate-high intensity exercise that involves resistance training and impact exercise versus posture and low intensity balance exercises. Women taking osteoporosis medication will be equally and randomly assigned to one of the exercise groups. There will be 23 participants per group and both exercise programs will be performed over a span of 6 months, twice weekly, for approximately 30-45 minutes per session. Investigators will measure sclerostin, a bone-related protein found in the blood, to see if there are any changes after 3 months of training. Higher levels of sclerostin may result in greater bone breakdown. It is expected that the moderate-high intensity exercise program will decrease sclerostin levels more than low intensity training. Further, changes in sclerostin levels during the 6-month exercise intervention will be explored. The effects of the exercise program on other bone markers in the blood, physical ability, and quality of life will be reported. The willingness of the participants to perform the exercise program and the safety of the exercises provided will also be assessed.

DETAILED DESCRIPTION:
Pharmacological and exercise interventions aimed to treat osteoporosis are typically examined separately. A common pharmacological treatment for osteoporosis involves antiresorptive medications, which has been previously shown to blunt the bone response to exercise. Many studies have shown that moderate-high intensity progressive resistance training (PRT) and impact exercise is required to stimulate bone. There are only two RCT studies that examined the effect of progressive resistance training or impact exercise on bone response in participants taking antiresorptive medications. One study showed that the combination of antiresorptive medications and resistance training did not increase bone mineral density (BMD) to a greater extent than medications alone in postmenopausal women. Another study demonstrated no additive effect of antiresorptive medications and progressive impact exercise on reducing bone turn over markers (BTMs) in postmenopausal women. However, there are currently no available studies that examine the effect of both progressive resistance training along with impact exercise on the bone response in women taking antiresorptive medications. Most exercise studies exclude people taking medications that affect bone, or are heterogeneous with respect to antiresorptive medication use. Further, there is little data on the safety of moderate-high intensity PRT and impact exercise in individuals at moderate or high risk for fracture.

The bone response to medications and exercise can be measured via the assessment of bone biomarkers present in the blood. For instance, sclerostin is a protein secreted by osteocytes and it can influence the bone remodeling process by inhibiting bone formation. Human genetic disorders deficient in sclerostin, such as sclerosteosis and Van Buchem's disease, have been associated with significant increases in bone mass. Therefore, decreasing sclerostin levels may be a potential treatment for people with low bone mass conditions. A case-control study demonstrated that postmenopausal women who adequately responded to bisphosphonates (e.g., did not experience a fracture while on treatment) had significantly lower serum sclerostin concentrations than those who experienced a fracture while taking bisphosphonates. There is also a link between sclerostin and exercise as a previous cross-sectional study reported an association between low serum sclerostin levels and increased physical activity duration. In addition, PRT and high impact exercise interventions have been shown to decrease sclerostin levels in healthy pre-menopausal women and thus may eventually increase bone mass or prevent bone loss. Therefore, changes in serum sclerostin levels can be used to provide insight regarding the bone response to antiresorptive medications as well as exercise.

Investigators plan to conduct a single-blinded parallel-group randomized controlled trial (RCT) with 1:1 allocation ratio to determine whether participants with low bone mass are able to adhere and safely perform PRT and impact exercises at an intensity that is hypothesized to stimulate bone. Specifically, the primary aim will be to determine the effects of moderate-high PRT and impact training on sclerostin in women on antiresorptive medication. The secondary aims are: a) to explore the effects of moderate-high PRT and impact training on BTMs [serum N-terminal procollagen of type I collagen (P1NP), C-terminal cross-linked of type I collagen (CTX), parathyroid hormone (PTH), Vitamin D and serum calcium], physical function and quality of life and body composition; b) to determine the feasibility of the intervention by assessing adherence, participant satisfaction with the intervention, and the acceptability of the attention control group; and c) to determine if there are any adverse events, including falls, fractures, or other adverse health outcomes attributable to the exercise intervention.

Investigators hypothesize that a moderate-to high PRT and impact exercise program will decrease sclerostin levels to a greater extent than the posture and balance exercise program. Further, it is hypothesized that PRT and impact exercise will result in more favourable improvements in other bone biomarkers, physical function, mobility, quality of life and body composition than the control group. Investigators hypothesize a low drop-out rate since both groups will be receiving the same level of attention throughout the study. Further, no adverse events attributable to exercise are expected. Kinesiologists who are Certified Exercise Physiologists will provide coaching on proper form, and will use appropriate progression of exercise intensity and volume.

Sample Size Estimation:

The sample size estimation was determined using data from a cross-sectional study that reported an association between low physical activity duration and high serum sclerostin levels. Women who engaged in less than 30 minutes of exercise per week had statistically significantly higher serum sclerostin levels than women who engaged in 60-120 minutes of physical activity per week (27.84 +/- 4.98 pmol/L vs. 21.64 +/- 6.21 pmol/L; p<0.0001, respectively). The study described used a manual ELISA® kit to assess sclerostin which is consistent with the current study protocol. Based on the study findings, to detect a difference in serum sclerostin of 6.2 pmol/L with a standard deviation of 1.23 pmol/L investigators will need 38 participants using an alpha level of 0.05 and a power of 90%. Investigators assumed a 20% attrition rate for the current study therefore the estimated sample size was increased to 46 participants.

Analyses:

The study protocol was prepared according to the Standard Protocol Items: Recommendations for Interventional Trial (SPIRIT) guidelines. Reporting will be consistent with Consolidated Standards of Reporting Trials (CONSORT) non-pharmacological trials extension. The proposed study protocol is summarized. Participant characteristics and outcomes that are considered continuous variables will be reported as mean +/- standard deviation or median and interquartile range. Categorical data will be reported as number (%). Analyses of the feasibility and safety of the exercise intervention will be descriptive. A participant flow diagram will be used to demonstrate the number of participants who were randomly assigned to each group, who completed the exercise training program and who were analyzed for each outcome. For each group, losses or exclusions after randomization will be recorded along with reasons. Intention-to-treat analysis will be performed and thus all participants will be included in the analysis and analysed according to the group to which they were randomized. Differences in outcome measures will be assessed using analysis of covariance (ANCOVA) while adjusting for baseline demographic and clinical characteristics (e.g., age, smoking status, physical activity level, dietary intake). Investigators will also perform sensitivity analysis to determine if participants with ≥80% adherence criteria to the exercise intervention experience greater benefits. At the end of the study, investigators will assess whether allocation concealment was maintained among the blinded research staff and whether participants were aware of the study hypothesis. Statistical significance will be set at p < or equal to 0.05. All data analysis will be conducted using the IBM Corporation Statistical Package for the Social Sciences (SPSS) version 24.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age AND
* Taking anti-resorptive medications for at least 12 months eg. risedronate (Actonel), alendronate (Fosamax, Fosavance), etidronate (Didronel, Didrocal), zoledronic acid (Aclasta, Reclast, Zometa), pamidronate (Aredia) and denosumab (Prolia, Xgeva).

Exclusion Criteria:

* Not able to communicate in English
* Already participating in structured progressive resistance exercise or impact training exercise program; presence of any progressive neurological disorders that can possibly prevent study completion; unable to stand or walk 10 m with or without gait aid; does not have the mental capacity to provide informed consent; have any contraindications to exercise as determined by a physician.
* Individuals that have had a fracture in the last 6 months need to have completed any immobilization (eg. casting) and post-fracture rehabilitation, and will need physician consent to participate in the study. Individuals with previous fractures (> 6 months ago) will not be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline Serum Sclerostin at 3 months and 6 months. | Baseline, 3-month and 6-month follow up.
  The primary outcome measure will be serum sclerostin. Venous blood samples will be taken by experienced phlebotomists between 8:00 and 10:00 am, after an overnight fast (8-12 hours). Participants will also be instructed to refrain from exercise for 48 hours prior to blood collection. An assessor who is blind to group allocation will measure sclerostin using ab221836 Human SOST SimpleStep ELISA® (Enzyme-Linked Immunosorbent Assay) supplied by Abcam (Abcam Inc., Toronto, Ontario, Canada).

SECONDARY OUTCOMES:
Descriptive Data - Demographic information | Baseline
  We will collect data such as demographic information including date of birth, race, formal education and marital status.
Descriptive Data - Medical History | Baseline
  Current and past medical history (including family history) will be collected including recent/past drug therapies and bone-related medications, reproductive history (e.g. age at menarche or menopause), past surgical history, falls risk (e.g. number of falls within the last 12 months) and fracture history, as well as current alcohol consumption and smoking status.
Descriptive Data - Physical Activity | Baseline
  Baseline physical activity will be assessed using a Bone-specific Physical activity Questionnaire (BPAQ), and by asking participants to wear accelerometers for one week prior to participating in the exercise program.
Descriptive Data - Dietary Intake | Baseline, 3-months, and 6-months
  To assess dietary energy, calcium and protein intake, participants will be asked to complete an Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool (Canada Version).
Other bone biomarkers - Serum P1NP | Baseline, 3-month and 6-month follow up.
  Serum P1NP will be be measured by the same single blinded assessor. P1NP will be measured using Human Total Procollagen Type I Intact N-Terminal Propeptide (TP1NP) ELISA Kit supplied by MyBioSource (MyBioSource Inc., San Diego, California, USA).
Other bone biomarkers - CTX | Baseline, 3-month and 6-month follow up.
  CTX will be measured in the blood by the same single blinded assessor. Beta-crosslaps CTX will be measured using Human beta-crosslaps (bCTx) ELISA Kit supplied by Cusabio (Cusabio Technology LLC, Houston, Texas, USA).
Other bone biomarkers - Parathyroid Hormone | Baseline, 3-month and 6-month follow up.
  PTH will be measured in the blood by the same single blinded assessor. Parathyroid hormone will be measured using ab230931 Human PTH SimpleStep ELISA® Kit supplied by Abcam (Abcam Inc., Toronto, Ontario, Canada).
Other bone biomarkers - Vitamin D | Baseline, 3-month and 6-month follow up.
  Vitamin D will be measured in the blood by the same single blinded assessor. Vitamin D will be measured using Human 25-Hydroxyvitamin D-1 Aplha Hydroxylase Mitochondrial (CYPB27B1) ELISA® Kit supplied by Cusabio (Cusabio Technology LLC, Houston, Texas, USA).
Other bone biomarkers - Calcium | Baseline, 3-month and 6-month follow up.
  Calcium will be measured in the blood by the same single blinded assessor. Calcium will be measured using ab112115 Calcium Quantification Kit - Red Fluorescence supplied by Abcam (Abcam Inc., Toronto, Ontario, Canada).
Physical function and mobility - 40 metre Fast-paced Walk | Baseline, 3-month and 6-month follow up.
  Physical function and mobility will be assessed using the 40 m fast-paced walk test. Time to complete test will be recorded.
Physical function and mobility - 30-second Sit-to-Stand Test | Baseline, 3-month and 6-month follow up.
  Physical function and mobility will be assessed using the 30-second sit-to-stand test. Number of sit-to-stand repetitions performed in 30 seconds will be recorded.
Physical function and mobility - 4-square Step Test | Baseline, 3-month and 6-month follow up.
  Physical function and mobility will be assessed using the 4-square step test. Time to complete test will be recorded.
Physical function and mobility - Stair Climb Test | Baseline, 3-month and 6-month follow up.
  Physical function and mobility will be assessed using the stair climb test. Time to complete test will be recorded.
Quality of Life - EQ-5D | Baseline, 3-month and 6-month follow up.
  The 5 level EuroQol EQ-5D instrument (EQ-5D-5L) will be used to assess the quality of life of the participants. The EQ-5D-5L instrument includes a descriptive system that is comprised of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores are coded from 11111 (no problems in all dimensions) to 55555 (extreme problems in all dimensions). A lower score is better. There is also a visual analogue scale that is used to measure the individuals self-rated overall health on a particular day. The visual analogue scale is scored from 0 (worst health imaginable) to 100 (best health imaginable).
Quality of Life - QUALEFFO-41 | Baseline, 3-month and 6-month follow up.
  The Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO-41) questionnaire will be used to assess quality of life of the participants. The QUALEFFO-41 questionnaire is specific to people with osteoporosis and includes the following domains: pain, activities of daily living, mobility, leisure and social activity, general health perception, and mental function. Scores range from 0-100, lower is better.
Bone Mineral Density | Baseline and 6 months.
  Certified technologists, blind to group allocation, will assess bone mineral density (g/cm2) at the spine (L1-L4) and femoral neck using a dual energy X-ray absorptiometry (DXA) scan (Hologic Inc, Bedford, MA).
Body Composition | Baseline and 6 months.
  Certified technologists, blind to group allocation, will assess body mass (kg) and use this to determine whole body fat- and bone-free lean mass (FBFM, in kg) and appendicular lean mass (ALM, in kg) and its index (ALMI) using a dual energy X-ray absorptiometry (DXA) scan (Hologic Inc, Bedford, MA).
Feasibility (Number of participants retained) | 6 months.
  Feasibility outcomes will include a record of the number of participants recruited and retained, and the acceptability of the attention control group (e.g., low dropout rate after randomization).
Feasibility (Adherence) | Through study, 6 months.
  The exercise trainers will be provided with an attendance sheet at every exercise session to monitor the number of exercise sessions participants attend to determine adherence.
Feasibility (Acceptability) | 6 months.
  We will conduct one exit interview to determine the participants' perspective on the intervention and control groups, and if they understood the purpose of the study.
Falls | Through study, up to 6 months
  Falls will be recorded using a prospective notification system to assess the number of falls, the number of fallers/non-fallers/frequent fallers and the fall rate. Participants will be asked weekly to report any falls that occurred outside of, and during, the exercise training program. Participants will be instructed to provide their weekly assessments to the exercise trainers when they attend their scheduled exercise sessions. Exercise trainers will check to ensure completion, confirm the date, injuries and hospitalization after a fall has been reported, and will follow-up with participants who have missing assessments.
Fractures | Through study, up to 6 months
  Participants will also be asked to report any new fractures or injuries, related or unrelated to the exercise training. Exercise trainers will complete an adverse event report to ascertain the cause and timing of any injuries. To verify fracture details, written consent will be obtained to abstract data from medical records.
Adverse Events | Through study, up to 6 months.
  According to Health Canada a serious adverse event is defined as ". . . an event (experience) or reaction is any untoward medical occurrence that at any dose (a) results in death, (b) is life-threatening, (c) requires inpatient hospitalization or prolongation of existing hospitalization, (d) results in persistent or significant disability/ incapacity, or (e) is a congenital anomaly/birth defect". Whereas a non-serious adverse event includes bone/limb pain, myalgia or muscle cramps (e.g. pain, cramps or aches), and injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Lora M Giangregorio, PhD, Principal Investigator — University of Waterloo, Schlegel-UW Research Institute for Aging
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

REFERENCES:
- [Background] Swift JM, Nilsson MI, Hogan HA, Sumner LR, Bloomfield SA. Simulated resistance training during hindlimb unloading abolishes disuse bone loss and maintains muscle strength. J Bone Miner Res. 2010 Mar;25(3):564-74. doi: 10.1359/jbmr.090811. PMID 19653816
- [Background] Chilibeck PD, Davison KS, Whiting SJ, Suzuki Y, Janzen CL, Peloso P. The effect of strength training combined with bisphosphonate (etidronate) therapy on bone mineral, lean tissue, and fat mass in postmenopausal women. Can J Physiol Pharmacol. 2002 Oct;80(10):941-50. doi: 10.1139/y02-126. PMID 12450060
- [Background] Uusi-Rasi K, Kannus P, Cheng S, Sievanen H, Pasanen M, Heinonen A, Nenonen A, Halleen J, Fuerst T, Genant H, Vuori I. Effect of alendronate and exercise on bone and physical performance of postmenopausal women: a randomized controlled trial. Bone. 2003 Jul;33(1):132-43. doi: 10.1016/s8756-3282(03)00082-6. PMID 12919708
- [Background] Martyn-St James M, Carroll S. A meta-analysis of impact exercise on postmenopausal bone loss: the case for mixed loading exercise programmes. Br J Sports Med. 2009 Dec;43(12):898-908. doi: 10.1136/bjsm.2008.052704. Epub 2008 Nov 3. PMID 18981037
- [Background] Basat H, Esmaeilzadeh S, Eskiyurt N. The effects of strengthening and high-impact exercises on bone metabolism and quality of life in postmenopausal women: a randomized controlled trial. J Back Musculoskelet Rehabil. 2013;26(4):427-35. doi: 10.3233/BMR-130402. PMID 23948830
- [Background] Erickson CR, Vukovich MD. Osteogenic index and changes in bone markers during a jump training program: a pilot study. Med Sci Sports Exerc. 2010 Aug;42(8):1485-92. doi: 10.1249/MSS.0b013e3181d0fa7a. PMID 20139789
- [Background] Watson S, Weeks B, Weis L, Harding A, Horan S, Beck B. High-Intensity Resistance and Impact Training Improves Bone Mineral Density and Physical Function in Postmenopausal Women With Osteopenia and Osteoporosis: The LIFTMOR Randomized Controlled Trial. J Bone Miner Res. 2019 Mar;34(3):572. doi: 10.1002/jbmr.3659. Epub 2019 Feb 25. No abstract available. PMID 30861219
- [Background] Watson SL, Weeks BK, Weis LJ, Horan SA, Beck BR. Heavy resistance training is safe and improves bone, function, and stature in postmenopausal women with low to very low bone mass: novel early findings from the LIFTMOR trial. Osteoporos Int. 2015 Dec;26(12):2889-94. doi: 10.1007/s00198-015-3263-2. Epub 2015 Aug 5. PMID 26243363
- [Background] Hamilton CJ, Swan VJ, Jamal SA. The effects of exercise and physical activity participation on bone mass and geometry in postmenopausal women: a systematic review of pQCT studies. Osteoporos Int. 2010 Jan;21(1):11-23. doi: 10.1007/s00198-009-0967-1. Epub 2009 Jun 6. PMID 19504035
- [Background] Beck BR, Daly RM, Singh MA, Taaffe DR. Exercise and Sports Science Australia (ESSA) position statement on exercise prescription for the prevention and management of osteoporosis. J Sci Med Sport. 2017 May;20(5):438-445. doi: 10.1016/j.jsams.2016.10.001. Epub 2016 Oct 31. PMID 27840033
- [Background] Kaastad TS, Nordsletten L, Narum S, Madsen JE, Haug E, Reikeras O. Training increases the in vivo fracture strength in osteoporotic bone. Protection by muscle contraction examined in rat tibiae. Acta Orthop Scand. 1996 Aug;67(4):371-6. doi: 10.3109/17453679609002334. PMID 8792742
- [Background] Howe TE, Shea B, Dawson LJ, Downie F, Murray A, Ross C, Harbour RT, Caldwell LM, Creed G. Exercise for preventing and treating osteoporosis in postmenopausal women. Cochrane Database Syst Rev. 2011 Jul 6;2011(7):CD000333. doi: 10.1002/14651858.CD000333.pub2. PMID 21735380
- [Background] Baron R, Rawadi G. Targeting the Wnt/beta-catenin pathway to regulate bone formation in the adult skeleton. Endocrinology. 2007 Jun;148(6):2635-43. doi: 10.1210/en.2007-0270. Epub 2007 Mar 29. PMID 17395698
- [Background] van Bezooijen RL, ten Dijke P, Papapoulos SE, Lowik CW. SOST/sclerostin, an osteocyte-derived negative regulator of bone formation. Cytokine Growth Factor Rev. 2005 Jun;16(3):319-27. doi: 10.1016/j.cytogfr.2005.02.005. PMID 15869900
- [Background] Moester MJ, Papapoulos SE, Lowik CW, van Bezooijen RL. Sclerostin: current knowledge and future perspectives. Calcif Tissue Int. 2010 Aug;87(2):99-107. doi: 10.1007/s00223-010-9372-1. Epub 2010 May 15. PMID 20473488
- [Background] Morales-Santana S, Diez-Perez A, Olmos JM, Nogues X, Sosa M, Diaz-Curiel M, Perez-Castrillon JL, Perez-Cano R, Torrijos A, Jodar E, Rio LD, Caeiro-Rey JR, Reyes-Garcia R, Garcia-Fontana B, Gonzalez-Macias J, Munoz-Torres M. Circulating sclerostin and estradiol levels are associated with inadequate response to bisphosphonates in postmenopausal women with osteoporosis. Maturitas. 2015 Dec;82(4):402-10. doi: 10.1016/j.maturitas.2015.08.007. Epub 2015 Aug 20. PMID 26358930
- [Background] Ardawi MS, Rouzi AA, Qari MH. Physical activity in relation to serum sclerostin, insulin-like growth factor-1, and bone turnover markers in healthy premenopausal women: a cross-sectional and a longitudinal study. J Clin Endocrinol Metab. 2012 Oct;97(10):3691-9. doi: 10.1210/jc.2011-3361. Epub 2012 Aug 3. PMID 22865898
- [Background] Vainionpaa A, Korpelainen R, Vaananen HK, Haapalahti J, Jamsa T, Leppaluoto J. Effect of impact exercise on bone metabolism. Osteoporos Int. 2009 Oct;20(10):1725-33. doi: 10.1007/s00198-009-0881-6. Epub 2009 Mar 5. PMID 19262975